CLINICAL TRIAL: NCT05663112
Title: Is Breast Massage Necessary to Find Sentinel Lymph Node After Isosulfan Blue Injection in Patients With Breast Cancer? A Prospective Randomized Study.
Brief Title: Is Breast Massage Necessary to Find Sentinel Lymph Node?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Sezgi Erel, Research assistant, MD, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.478.486
Record Dates: First submitted 2021-12-22; First posted 2022-12-23 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Sentinel Lymph Node; Breast Cancer
Keywords: breast cancer; isosulfan blue; massage; sentinel lymph node; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: This research is a prospective randomized study. Patients will be randomized by number-drawing method. Patients with BMI>30 and age>65 will be equally distributed to the experimental and active comparator arms. Under general anesthesia patients will be injected with 5 ml of isosulfan blue into the subareolar region. In one group, breast massage will be applied for 5 minutes. In the other group no massage will be applied. Surgical team will wait for a duration of 5 minutes for the self distribution of the blue dye.
Masking Description: not necessary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm with massage (Active Comparator): 5 ml of isosulfan blue will be injected into the subareolar region. 5-minutes massage will be applied.
  Drug: Isosulfan Blue 5 ml
  Interventions: Procedure: Sentinel lymph node biopsy; Procedure: Breast massage; Procedure: Blue dye injection
- Arm without massage (Experimental): 5 ml of isosulfan blue will be injected into the subareolar region. No massage will be applied.
  Drug: Isosulfan Blue 5 ml
  Interventions: Procedure: Sentinel lymph node biopsy; Procedure: Blue dye injection

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy — Sentinel lymph node biopsy will be performed.
Procedure: Breast massage — Breast massage will be performed for a duration of 5 minutes.
  Arms: Arm with massage
Procedure: Blue dye injection — Isosulfan blue dye will be injected in the subareolar region of the breast

SUMMARY:
Sentinel lymph node biopsy is important for staging in patients with breast cancer and changes the way of surgery. One of the most commonly used methods to find the sentinel lymph node during surgery is to apply blue dye around the areola and then search for the sentinel lymph node. Breast massage is recommended following administration of the blue dye. However, the necessity of this massage is controversial. In this study, investigators will try to find out whether massage of the breast after blue dye injection has any positive effect on finding the sentinel lymph node.

DETAILED DESCRIPTION:
This research is a prospective randomized study. Patients will be randomized by number-drawing method. Patients with BMI>30 and age>65 will be equally distributed to the experimental and active comparator arms. Under general anesthesia patients will be injected with 5 ml of isosulfan blue into the subareolar region. In one group, breast massage will be applied for 5 minutes. In the other group no massage will be applied. Surgical team will wait for a duration of 5 minutes for the self distribution of the blue dye.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of breast cancer by biopsy
* participants voluntarily participated in the clinical trial and signed informed consent

Exclusion Criteria:

* had previous sentinel lymph node biopsy or axillary surgery
* had neoadjuvant chemotherapy
* had clinical hints of axillary lymph node metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Sentinel lymph node detection rate | 2 weeks
  Participants will be followed until the pathology report is finalized

CONTACTS AND LOCATIONS:
Overall Officials: Teoman Coskun, Prof., Study Director — Celal Bayar University Department of General Surgery
Locations (1):
- Celal Bayar University, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data sharing will not contribute to other researchers

REFERENCES:
- [Result] Shenoy V, Ravichandran D, Ralphs DN. Is massage following dye injection necessary in sentinel node biopsy in breast cancer? Breast. 2002 Jun;11(3):273-4. doi: 10.1054/brst.2002.0415. PMID 14965682
- [Result] Bass SS, Cox CE, Salud CJ, Lyman GH, McCann C, Dupont E, Berman C, Reintgen DS. The effects of postinjection massage on the sensitivity of lymphatic mapping in breast cancer. J Am Coll Surg. 2001 Jan;192(1):9-16. doi: 10.1016/s1072-7515(00)00771-7. PMID 11192930
- [Result] Diaz NM, Vrcel V, Centeno BA, Muro-Cacho C. Modes of benign mechanical transport of breast epithelial cells to axillary lymph nodes. Adv Anat Pathol. 2005 Jan;12(1):7-9. doi: 10.1097/01.pap.0000151267.34438.a1. PMID 15614159
- See also: Is massage following dye injection necessary in sentinel node biopsy in breast cancer? — http://pubmed.ncbi.nlm.nih.gov/14965682/
- See also: The Effects of Postinjection Massage on the Sensitivity of Lymphatic Mapping in Breast Cancer — http://pubmed.ncbi.nlm.nih.gov/11192930/
- See also: Modes of Benign Mechanical Transport of Breast Epithelial Cells to Axillary Lymph Nodes — http://pubmed.ncbi.nlm.nih.gov/15614159/